CLINICAL TRIAL: NCT00606450
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Dose Comparison Study of CC-10004 in Subjects With Moderate-to-Severe Plaque-Type Psoriasis
Brief Title: Double-Blind, Randomized, Placebo-controlled Comparison of CC-10004 in Subjects With Moderate to Severe Plaque Type Psoriasis
Acronym: PSOR-003
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CC-10004-PSOR-003
Record Dates: First submitted 2008-01-22; First posted 2008-02-04 (Estimated); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Psoriasis
Keywords: plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 20 mg Apremilast daily (Experimental): 20 mg of CC-10004 daily
  Interventions: Drug: CC-10004
- 20mg Apremilast twice daily (Experimental): CC-10004 twice daily
  Interventions: Drug: CC-10004
- Placebo (Placebo Comparator): Placebo arm
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: CC-10004 — 20 mg CC-10004 taken 1 time per day for 12 weeks
  Other Names: Apremilast
  Arms: 20 mg Apremilast daily
Drug: CC-10004 — 20 mg of CC-10004 taken 2 times per day for 12 weeks
  Other Names: Apremilast
  Arms: 20mg Apremilast twice daily
Drug: Placebo — matching placebo taken either 1 or 2 times per day for 12 weeks
  Arms: Placebo

SUMMARY:
There is an unmet medical need for safe, effective oral therapy for moderate-to-severe psoriasis. CC-10004 will be evaluated in a controlled setting of a clinical study. The information obtained from the study will aid in the design of future clinical trials and to establish the safety and efficacy of CC-10004.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and voluntarily sign and informed consent form
* Must be in good health as judged by the investigator
* Must be able to adhere to the study visit schedule and other protocol requirements
* Must have greater than or equal to a 6 month history of moderate-to-severe plaque-type psoriasis
* Must have a Psoriasis Area and Severity Index (PASI) score greater than or equal to 10 and Body Surface Area (BSA) greater than or equal to 10%
* Must meet specific laboratory criteria
* Must be a candidate for photo/systemic therapy
* Women of childbearing potential must have a negative pregnancy test

Exclusion Criteria:

* Must not have clinically significant underlying disease processes
* Must not be pregnant or lactating females
* Must not have any condition, including lab abnormalities, which places the subject at unacceptable risk if the subject were to participate in the study or confounds the ability to interpret data from the study
* Must not have a history of active mycobacterium tuberculosis infection within 3 years prior to the screening visit
* Must not have a history of incompletely treated active of latent mycobacterium tuberculosis infection
* Must not have a know history of exposure to an infectious case of mycobacterium tuberculosis within 2 years prior to the screening visit
* Must not be an immigrant form a high-incidence country for mycobacterium tuberculosis disease within 2 years prior to the screening visit
* Must not have current erythrodermic, guttate, or pustular psoriasis
* Must not have a clinical history of failure to adequately respond to treatment in the investigator's opinion to one or more treatment courses of cyclosporine or the following biologic therapies: alefacept, etanercept, efalizumab, infliximab or adalimumab
* Must not use topical therapy within 14 days of randomization
* Must not use systemic therapy for psoriasis within 28 days of randomization
* Must not use phototherapy within 28 days of randomization
* Must not use adalimumab or infliximab within 3 months of randomization
* Must not use etanercept or efalizumab within 56 days of randomization
* Must not use alefacept within 6 months of randomization

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2006-04-01 (Actual); Primary Completion 2007-02-01 (Actual); Study Completion 2007-05-01 (Actual)

PRIMARY OUTCOMES:
To compare the clinical efficacy of 2 oral doses of CC-10004 with placebo when taken for 12 weeks in subjects with moderate-to-severe plaque-type psoriasis | 12 weeks

SECONDARY OUTCOMES:
To evaluate the safety of CC-10004 compared with placebo in subjects with moderate-to-severe placque-type psoriasis | 12 weeks
To evaluate the effects of CC-10004 compared to placebo on the quality of life in subjects with moderate-to-severe plaque-type psoriasis. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen
Locations (31):
- Canada (11):
  - Division of Dermatology and Cutaneous Science, Edmonton, Alberta
  - Division of Dermatology, Vancouver, British Columbia
  - Duronder C.P. Inc, Moncton, New Brunswick
  - Eastern Canada Cutaneous Research Associates, Halifax, Nova Scotia
  - Ultranova Skincare, Barrie, Ontario
  - Dermatrials Research, Hamilton, Ontario
  - The Lynde Center for Dermatology, Markham, Ontario
  - North Bay Dermatology Centre, North Bay, Ontario
  - K. Papp Clinical Research, Waterloo, Ontario
  - Innovaderm, Montreal, Quebec
  - Dr Yves Poulin, Québec, Quebec
- Czechia (5):
  - Department of Dermatology, Brno
  - Department of Dermatology, Hradec Králové
  - Department of Dermatovererology, Olomouc
  - Department of Dermatovererology, Prague
  - Depart of Dermatology, Ústí nad Labem
- Germany (15):
  - Celgene Clinical Site, Ausburg
  - Celgene Clinical Site, Berlin
  - Department of Dermatologie and Venerology, Dresden
  - Department of Dermatology and Venerology, Frankfurt am Main
  - Celgene Clinical Site, Hamburg
  - Celgene Clinical Site, Heidelberg
  - Celgene Clinical Site, Herborn
  - Celgene Clinical Site, Homburg
  - Celgene Clinical Site, Leipzig
  - Celgene Clinical Site, Mannheim
  - Celgene Clinical Site, Münster
  - Celgene Clinical Site, Salzwedel
  - Celgene Clinical Site, Schwerin
  - Celgene Clinical Site, Wiesbaden
  - Celgene Clinical Site, Würzburg

REFERENCES:
- [Background] Papp KA, Kaufmann R, Thaci D, Hu C, Sutherland D, Rohane P. Efficacy and safety of apremilast in subjects with moderate to severe plaque psoriasis: results from a phase II, multicenter, randomized, double-blind, placebo-controlled, parallel-group, dose-comparison study. J Eur Acad Dermatol Venereol. 2013 Mar;27(3):e376-83. doi: 10.1111/j.1468-3083.2012.04716.x. Epub 2012 Oct 3. PMID 23030767